CLINICAL TRIAL: NCT02623946
Title: Motor Evoked Potentials as a Biomarker in Alemtuzumab Treated Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Clinique Neuro-Outaouais (Other)
Collaborators: CogState Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Francois Jacques, neurologist, Clinique Neuro-Outaouais
Other Study IDs: CNO-004
Record Dates: First submitted 2015-11-30; First posted 2015-12-08 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis
Keywords: motor evoked potentials
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Design:

Phase 4, pilot, single center, observational study. MEP's will be obtained twice, two weeks apart at baseline and every 6 months for 36 months (total of 14 sessions of MEP's)

MEP's will include:

1. Onset latencies and CMCT to bilateral abductor pollicis brevis and tibialis anterior muscles
2. MEP amplitudes and the ratio of the central to peripherally obtained motor amplitudes (MEP-M ratio) to bilateral abductor pollicis brevis and tibialis anterior muscles Clinical measures (EDSS, MEP's, T25FWT, 6MWT, 9HPT) will be obtained at baseline and every 6 months for 36 months.

Study location: Single center in Canada

Study Objectives:

Primary: To evaluate the reliability of MEP's in Alemtuzumab treated MS patients over a 36 month period.

Secondary: To determine the degree of correlation between MEP's and presently used clinical measures of efficacy (EDSS, 6MWT, T25FWT, 9HPT) and to determine if MEP's can predict who will require a third cycle of Alemtuzumab.

DETAILED DESCRIPTION:
Alemtuzumab pivotal studies have shown robust effect on relapse rate and MRI parametric. The effect on disease progression did not however reach statistical significance in CARE MS I Clinical trials, especially in the progressive forms of Multiple Sclerosis (MS) have been greatly hampered by the insensitivity of the Expanded Disability Status Scale (EDSS) especially at either ends of the scale. Other more recently introduced clinical scales such the timed 25 foot walk test (T25FWT), six minute walk test (6MWT) or the 9-hole peg test (9HPT) also lack in sensitivity and reliability. A validated, sensitive and reliable biomarker for disability progression or regression would greatly help clinical research in MS. Such a biomarker could also help in evaluating if and when patients would require retreatments with Alemtuzumab.

Motor evoked potentials (MEP's) measures the integrity and function of corticospinal tracts. The procedure uses an electromagnet to induce directly or via interneurons a small depolarizing current in the axon hillock of large pyramidal neurons in the motor cortex. A subsequent motor response can then be measured in the targeted limb muscle. The amplitude and latency of such response can be measured giving an indication of the conduction integrity of the corticospinal tracts (CST) from the cortex to the limb. MEP's are able to detect perhaps even before clinical measures, evidence of CST involvement and deterioration through increased central motor conduction time and/or reduced ratio of centrally elicited MEP amplitude to peripherally elicited compound motor amplitude potential (CMAP).

MEP's have been studied in a variety of pathologies involving CST's. MEP's have in patients with cervical spondylosis as well as with patients with amyotrophic lateral sclerosis, shown to being more sensitive than clinical examination in detecting CST involvement. MEP's have been shown in MS to correlate with EDSS scores. In studies looking at spinal cord injury patients MEP's were able to demonstrate an improvement in central motor conduction time (CMCT) induced by extended release fampridine.

The main critique of MEP's has been as in all electrophysiological tests one of high intra-patient variability which can be compounded by non-standardized techniques between centers. Newer MEP techniques using neuro-navigation, standardized facilitation techniques and choosing the best of three responses can significantly reduce the inherent variability of obtained values. We believe that with such techniques MEP's can become a useful surrogate biomarker in clinical trials of MS. The latter however needs to be validated in a prospective manner.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS (McDonald criteria) and of age 18 and older;
* Subjects who meet the prescribing criteria for Alemtuzumab as per product monograph;
* An EDSS of 5.0 or less and a pyramidal system functional assessment score of 2 or greater;
* Subject who have received the first cycle of Alemtuzumab within the last 3 months.

Exclusion Criteria:

* Subjects who have begun using extended release Fampridine within 2 months of study baseline visit (Patient on a stable dose of extended release Fampridine for more than 2 months can enter the study);
* Subjects with MSSS (Multiple Sclerosis Severity Score) less than 4.0;
* Subject with other medical conditions that involve the CST's;
* Any other condition that would preclude them from undergoing the MEP's and/or MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MacDonald criteria (2005) multiple sclerosis presently being treated with Alemtuzumab.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
intrapatient correlation coefficient of MEP's | obtained between two assessments done two weeks apart
  to measure within subject correlation a two-way fixed Intraclass Correlation (ICC) will be calculated for each of 10 participants across sessions measured two weeks apart. The ICC will provide an estimate of the variance of each individual's motor evoked potentials at each paired time point.

SECONDARY OUTCOMES:
Correlation coefficient between the changes from baseline MEP results and clinical measures (EDSS, 6MW, T25FWT, 9HPT) | obtained every 6 months for 36 months
  to measure the relationship between MEP change scores and the change scores of the clinical measures, several correlations will be run across 6 months intervals over the 36 month period. The corrrelation between the individual changes in MEP results and the propensity to require a third cycle of alemtuzumab will also be calcutlated.
Correlation between the change in the conduction index and the change in clincal measures | obtained at baseline and every 6 months over 36 months
  to measure the correlation betwen the conduction index results and the clinical measures and the change in the conduction index over time and the change in the clinical measures over the 36month period.

CONTACTS AND LOCATIONS:
Overall Officials: Francois H Jacques, MD, Principal Investigator — Clinic Neuro-Outaouais; Director
Locations (1):
- Clinique Neuro-Outaouais, Gatineau, Quebec, Canada

REFERENCES:
- [Derived] Jacques FH, Apedaile BE, Danis I, Sikati-Foko V, Lecompte M, Fortin J. Motor Evoked Potential-A Pilot Study Looking at Reliability and Clinical Correlations in Multiple Sclerosis. J Clin Neurophysiol. 2024 May 1;41(4):357-364. doi: 10.1097/WNP.0000000000001003. Epub 2023 Mar 21. PMID 36943437